CLINICAL TRIAL: NCT02961491
Title: Expanded Access Program of AZEDRA (Ultratrace Iobenguane I131) in Subjects With Malignant Relapsed/Refractory Pheochromocytoma/Paraganglioma: A Sub-study of Protocol MIP-IB12B
Brief Title: Expanded Access Program of Ultratrace Iobenguane I131 for Malignant Relapsed/Refractory Pheochromocytoma/Paraganglioma
Status: Approved for marketing | Type: Expanded Access
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MIP-IB12B-EAP
Record Dates: First submitted 2016-11-08; First posted 2016-11-11 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Pheochromocytoma; Paraganglioma
Keywords: MIBG; Azedra; Rare neuroendocrine tumors; Iobenguane I 131; Progenics
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma | interventions — 3-Iodobenzylguanidine

INTERVENTIONS:
Drug: Ultratrace Iobenguane I131 — Subjects will receive a dosimetry dose of AZEDRA and will undergo 3 whole body scans. If the scans indicate tumor avidity for AZEDRA, the subjects will receive up to 2 therapeutic doses of AZEDRA each at 500 mCi (or 8 mCi/kg, for subjects weighing 62.5 kg or less) approximately 90 days apart.
  Other Names: Azedra; MIBG

SUMMARY:
The purpose of this sub-study is to provide expanded access of AZEDRA (Ultratrace Iobenguane I 131) and to evaluate the safety and tolerability of AZEDRA in subjects with iobenguane-avid malignant and/or recurrent pheochromocytoma/paraganglioma (PPGL).

DETAILED DESCRIPTION:
MIP-IB12B, the pivotal phase 2 study evaluating efficacy and safety of AZEDRA in patients with malignant relapsed/refractory PPGL, has completed its anticipated enrollment. The purpose of this sub-study, MIP-IB12B-EAP, is to provide expanded access to AZEDRA for newly enrolled subjects with iobenguane-avid metastatic and/or recurrent PPGL and to collect additional safety data.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent/assent and comply with protocol requirements
* Documented diagnosis of either pheochromocytoma or paraganglioma that was confirmed by histology or other supportive data (e.g. abnormal MIBG diagnostic study or elevated tumor markers)
* Ineligible for curative surgery for PPGL
* Failed a prior therapy for PPGL or have no alternative indicated therapy available
* Have definitive tumor avidity confirmed by the AZEDRA dosimetry dose
* Life expectancy of at least 6 months per physician

Exclusion Criteria:

* Pregnant or nursing females
* Men or women of childbearing potential and unwilling to use a medically acceptable form of contraception from time of consent until 6 months following last therapeutic dose of AZEDRA
* Active CNS lesions by CT/MRI within 3 months of informed consent
* NYHA class IV heart failure, unstable angina pectoris or clinically significant cardiac arrhythmia that poses a risk of syncope or cardiac arrest
* Prior systemic radiotherapy resulting in marrow toxicity within 3 months of first AZEDRA therapeutic dose
* Prior iobenguane I 131 therapeutic exposure within 12 weeks of the first planned therapeutic dose
* Prior administration of whole-body radiation therapy within 12 weeks of the first planned therapeutic dose
* Prior external beam radiotherapy to > 25% of bone marrow
* Prior chemotherapy or investigational compound and/or device within 30 days of the dosimetry dose
* Other active malignancy requiring additional treatment except for superficial cutaneous neoplasms
* Karnofsky Performance Status < 60
* Clinically significant laboratory abnormalities prior to dosing as listed in the protocol (such as blood count abnormalities, liver enzyme abnormalities, and renal dysfunction)
* Medical history of AIDS/HIV+
* Active chronic alcohol abuse, chronic liver disease (not including liver metastases), hepatitis A, B, or C
* Known allergy to iobenguane that has required medical intervention
* Receiving a medication which inhibits tumor uptake of iobenguane I 131
* Any other condition, that in the opinion of the investigator, may compromise the safety or compliance of the subject

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Iowa, Iowa City, Iowa
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas